CLINICAL TRIAL: NCT02763033
Title: Dietary Manipulation of the Microbiome-metabolomic Axis for Mitigating GVHD in Allo HCT Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UMCC 2016.029; HUM00112318 (Other: The University of Michigan); P01HL149633 (NIH)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bob's Red Mill® (Experimental): Patients will follow the standard BMT (bone marrow transplant) diet and add potato-starch produced by Bob's Red Mill® beginning on day -7 and continuing through day +100.Patients will consume 20 g of Bob's Red Mill®, Potato-based dietary starch, orally twice daily.
  Initially, subjects will take 20g daily for first three days prior to increasing dose to 20 g BID.
  Interventions: Drug: Bob's Red Mill®; Other: Starch Placebo
- Starch Placebo (Placebo Comparator): Patients will receive an iso-caloric, non-resistant starch placebo.
  Interventions: Other: Starch Placebo

INTERVENTIONS:
Drug: Bob's Red Mill® — Standard bone marrow transplant (BMT) diet + potato-based starch
  Arms: Bob's Red Mill®
Other: Starch Placebo — Standard bone marrow transplant (BMT) diet + corn-based starch

SUMMARY:
Investigators are evaluating the feasibility, safety and early efficacy of administering a commercially available dietary supplement containing potato-based resistant starch to subjects undergoing allogeneic SCT (stem cell transplant). The intervention will begin immediately prior to the conditioning phase and continue through day 100. Investigators hypothesize that short term administration of a resistant starch is capable of increasing levels of butyrate within the intestine that will reduce rates of acute GVHD (Graft-Versus-Host Disease).

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing matched related and matched unrelated full intensity allogeneic HSCT.
* Age ≥ 18 years for the feasibility phase. Age ≥10 years old AND ≥50 kg for the phase II portion.
* Karnofsky >70%, (Karnofsky Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 100 where 100 is "perfect" health and 0 is death.)
* Subjects must be able to swallow capsules/tablets
* Ability to understand and the willingness to sign a written informed consent
* Willingness to consent / co-enroll on BMT long term follow up study or HUM00043287 (UMCC2001-0234)
* Availability of an HLA matched related or matched unrelated donor

Exclusion Criteria:

* Patients with inflammatory bowel disease.
* Patients with a history of gastric bypass surgery.
* Patients with active Clostridium difficile infection at the time of study enrollment. Active infection is defined as a stool sample positive for Clostridium difficile toxin via EIA (enzyme immunoassay) and either symptoms (frequent loose stools) OR imaging findings consistent with toxic megacolon.
* Patients actively enrolled on any other GVHD prevention trial.
* Any physical or psychological condition that, in the opinion of the investigator, would post unacceptable risk to the patient or raise concern that the patient would not comply with protocol procedures.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade II-IV GVHD | Day 100
  The incidence of grade II, III and IV GVHD (Graft Versus Host Disease) as documented on day 100
  Grade II: Rash 25-50% of Body Surface Area (BSA), Bilirubin 3.1-6mg/dL, adult stool output 1000-1500mL/day or child 20-30mL/kg/day.
  Grade III: Rash greater than 50% BSA, bilirubin 6.1-15mg/dL, adult stool output greater than 1500mL/day or child stool output greater than 30mL/kg/day
  Grade IV: generalized erythroderma plus bullous formation and desquamation greater than 5% BSA, bilirubin greater than 15mg/dL, severe abdominal pain with or without ileus, or grossly bloody stool.

CONTACTS AND LOCATIONS:
Overall Officials: Mary M Riwes, D.O., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Riwes MM, Golob JL, Magenau J, Shan M, Dick G, Braun T, Schmidt TM, Pawarode A, Anand S, Ghosh M, Maciejewski J, King D, Choi S, Yanik G, Geer M, Hillman E, Lyssiotis CA, Tewari M, Reddy P. Feasibility of a dietary intervention to modify gut microbial metabolism in patients with hematopoietic stem cell transplantation. Nat Med. 2023 Nov;29(11):2805-2813. doi: 10.1038/s41591-023-02587-y. Epub 2023 Oct 19. PMID 37857710
- [Derived] Lakshmanan AP, Deola S, Terranegra A. The Promise of Precision Nutrition for Modulation of the Gut Microbiota as a Novel Therapeutic Approach to Acute Graft-versus-host Disease. Transplantation. 2023 Dec 1;107(12):2497-2509. doi: 10.1097/TP.0000000000004629. Epub 2023 May 16. PMID 37189240